CLINICAL TRIAL: NCT04086069
Title: Effect of Sit-to-stand Trainer in Patients With Unilateral Lower Limb Amputation on the Ability of Independent Standing up
Brief Title: Sit-to-stand Trainer in Patients After Lower Limb Amputation
Acronym: STSTrainer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Main clinician cancelled collaboration for personal reasons.
Sponsor: University Rehabilitation Institute, Republic of Slovenia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: URIS201903
Record Dates: First submitted 2019-09-05; First posted 2019-09-11 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Lower Limb Amputation
Keywords: unilateral lower-lim amputation; sit-to-stand trainer device; 30-Second Chair Stand Test; kinesiological analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Training+Sit-to-stand trainer (Experimental): Training using a sit-to-stand trainer device in addition to standard training of standing-up with the help of a physiotherapist
  Interventions: Device: Sit-to-stand trainer
- Standard Training (No Intervention): Standard training of standing-up with the help of a physiotherapist

INTERVENTIONS:
Device: Sit-to-stand trainer — The sit-to-stand trainer device is an exoskeleton that enables standing-up movement resembling the movement of a healthy person. It consists of three sub-systems: a foldable chair, a lever for body orientation and a triggering mechanism. It includes a support for feet with adjustable height. The device offers partial support to the patient while standing up. The patient will exercise with the device for 10 sessions (one per day), standing up for up to 30 times per session.
  Arms: Standard Training+Sit-to-stand trainer

SUMMARY:
The study will include rehabilitation inpatients after unilateral lower limb amputation who are candidates for walking with a prosthesis. Those in the experimental group will receive training using a sit-to-stand trainer device in addition to standard training of standing-up with the help of a physiotherapist. Those in the control group will only receive the standard training. The effects of the rehabilitation programme will be assessed using the 30-Second Chair Stand Test before the start of the training and after 10 days of training. For the first five patients from each group who will be able to stand up with the use of hands, detailed kinesiological analysis of standing-up pattern will be performed.

ELIGIBILITY:
Inclusion Criteria:

* unilateral lower-limb amputation
* candidate for walking with a prosthesis
* Montreal Cognitive Assessment (MoCA) test score 26 or more

Exclusion Criteria:

* associated neurological or orthopaedic disease
* amputation caused by cancer or injury
* BMI below 18.5 or above 30

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Change in 30-Second Chair Stand Test | Change from day 0 to day 10
  The test measures the number of times the participant is able to stand and return to a seated position in a chair in 30 seconds.

SECONDARY OUTCOMES:
Standing-up pattern | On day 10 after the last training session
  Detailed qualitative kinesiological analysis Will be performed to determine the standing-up pattern.

OTHER OUTCOMES:
Berg Balance Scale | On day 10 after the last training session
  The scale measures functional balance. The participants are asked to perform 14 tasks frequently used in daily life activities. The highest possible score is 56 points. A higher score indicates better balance.
6-Minute Walk Test | On day 10 after the last training session
  The test measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. Longer distance indicates better functional capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Helena Burger, MD, PhD, Principal Investigator — University Rehabilitation Institute, Republic of Slovenia
Locations (1):
- University Rehabilitation Institute, Republic of Slovenia, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] B Aledi L, Flumignan CD, Trevisani VF, Miranda F Jr. Interventions for motor rehabilitation in people with transtibial amputation due to peripheral arterial disease or diabetes. Cochrane Database Syst Rev. 2023 Jun 5;6(6):CD013711. doi: 10.1002/14651858.CD013711.pub2. PMID 37276273